CLINICAL TRIAL: NCT05645796
Title: Improved Chest CT Diagnostic and Contrast Medium Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Safora Johansen, Associate professor, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2016/674
Record Dates: First submitted 2022-11-28; First posted 2022-12-12 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-12

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: Two groups receiving contrast medium based on different approaches are included and compared with each other
Who Masked: Participant
Masking Description: Patients receiving contrast enhanced chest CT examination
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed group (Active Comparator): They received a fixed amount of contrast media prior to CT scan
  Interventions: Other: Adopted contrast media amount by using different approaches
- body composition tailored group (Active Comparator): They received a body tailored amount of contrast media prior to CT scan
  Interventions: Other: Adopted contrast media amount by using different approaches

INTERVENTIONS:
Other: Adopted contrast media amount by using different approaches — Using different contrast media approaches recommended by literature to explore the impact on the contrast enhancement in chest CT

SUMMARY:
Investigation of impact of using different CM approaches on contrast enhancement in chest Ct examinations - A prospective study

DETAILED DESCRIPTION:
Continuing advances in computed tomography (CT) in the past decades such as short scanning times with multi-detector CT (MDCT) requires contrast medium (CM) administration to be precisely planned to ensure a diagnostically accurate CT scans. To improve the chest CT diagnostic, the contrast enhancement in the thoracic vessels shoulde be increased.

The most important patient-related factors affecting the magnitude of vascular and parenchymal contrast enhancement are body weight. Historical practice has been to use a fixed volume of CM independent of body weight. Research has shown a clear relationship between vessel enhancement and patient weight, and that fixed CM volume technique is inappropriate, as smaller patients may receive excessive volume, and larger patients insufficient volume resulting in reduced image quality and poor diagnostic. In addition, excess CM can result in contrast induced adverse effects and nephropathy. To overcome these problems, it is essential to adjust the CM volume to the patient's total body weight and body composition. This adjustment can be done in different ways. The aim of this study is to identify which weight/body tailored CM administration is the best replacement for fixed CM administration in chest CT. The cost and procedure time will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing chest CT examination between August 2019 and September 2021
* age > 18 years

Exclusion Criteria:

* hemodynamic instability
* cardiac failure
* pacemaker
* renal insufficiency (estimated glomerular filtration rate <30 mL/min/1.73 m2)
* contraindications to contrast enhanced CT
* age < 18 years

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Contrast medium protocols in routine chest CT - A survey study | 15 months
  survey of what kind of contrast medium approaches are used in European hospitals

CONTACTS AND LOCATIONS:
Overall Officials: Safora F Johansen, PhD, Study Director — Oslo Metropolitan University
Locations (1):
- OsloMet University, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henning MK, Gunn C, Arenas-Jimenez J, Johansen S. Strategies for calculating contrast media dose for chest CT. Eur Radiol Exp. 2023 Jun 12;7(1):29. doi: 10.1186/s41747-023-00345-w. PMID 37303003